CLINICAL TRIAL: NCT00879476
Title: An Open Label, Balanced, Randomised, Two-Treatment, Two-Period, Two-Sequence, Single-Dose, Crossover, Bioavailability Study Comparing Ramipril 10 mg Capsules of OHM Laboratories Inc (a Subsidiary of Ranbaxy Pharmaceuticals Inc) With ALTACE® 10 mg Capsules (Containing Ramipril 10 mg) of King Pharmaceuticals Inc, in Healthy, Adult, Male Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Ramipril 10 mg Capsules Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 245_RAMIP_06
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Bioequivalence ramipril fasting condition
MeSH Terms: interventions — Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ramipril capsules 10 mg (containing Ramipril 10 mg)of of OHM Laboratories Inc., USA (a subsidiary of Ranbaxy Pharmaceuticals Inc), USA
  Interventions: Drug: Ramipril 10mg capsules
- 2 (Active Comparator): ALTACE® capsule 10 mg (containing Ramipril 10 mg)of King Pharmaceuticals Inc., Bristol, TN 37620, USA
  Interventions: Drug: Ramipril 10mg capsules

INTERVENTIONS:
Drug: Ramipril 10mg capsules

SUMMARY:
The study was conducted as an open label, balanced, randomized, two-treatment, two-period, two-sequence, single-dose, crossover bioavailability study comparing Ramipril capsules 10 mg of OHM Laboratories Inc., USA with ALTACE® (ramipril) capsule 10 mg manufactured by King Pharmaceuticals Inc., Bristol, TN 37620, USA in healthy, adult, male, human subjects under fasting condition.

DETAILED DESCRIPTION:
Following an overnight fast of at least 10 hour, a single oral dose of ramipril 10 mg capsule was administered during each period of the study, along with 240 mL of drinking water at ambient temperature, under low light condition and supervision of trained study personnel.

A total of sixty-eight (68) subjects were enrolled into the study, to be administered a single oral dose of the test or reference formulation of ramipril 10 mg capsule according to a randomization schedule. Two subjects (subject numbers 01 and 06) were withdrawn from the study in period I and subject number 02 did not report for period II.

Sixty-five (65) subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Were in the age range of 18-45 years.
2. Were neither overweight nor underweight for the corresponding height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Had voluntarily given written informed consent to participate in this study.
4. Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

1. Hypersensitivity or allergy to ramipril or related group of drugs.
2. Subject who had sitting systolic blood pressure of less than 90 mmHg or >140 mmHg and diastolic blood pressure of less than 60 mmHg or > 90 mm Hg at screening
3. History of hypertension, hypotension, angina, myocardial infarction or angioedema.
4. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
5. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes, glaucoma or angioedema due to any cause.
6. History of any psychiatric illness which might impair the ability to provide written informed consent.
7. Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
8. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
9. Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
10. Presence of values which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
11. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), glucose (positive) or protein (positive).
12. Clinically abnormal ECG or Chest X-ray.
13. Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
14. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit -equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
15. Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
16. Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
17. Subjects who, through completion of this study, would have had donated and/or lost more than 350 mL of blood in the past month.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence evaluation of Ranbaxy Ramipril 10mg Capsules under fasting conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Clinical Pharmacology Unit, Ranbaxy Laboratories Limited, Noida, Uttar Pradesh, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html